CLINICAL TRIAL: NCT00864201
Title: A Pilot Study to Evaluate the Effect of Bosentan in Patients With Exercise Induced Pulmonary Arterial Hypertension Associated With Connective Tissue Disease
Brief Title: A Study to Evaluate the Use of Bosentan in Patients With Exercise Induced Pulmonary Arterial Hypertension Associated With Connective Tissue Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Actelion (Industry)
Responsible Party: Dr. Christine Bradley, Victoria Medical Centre
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAH-CTD-2007
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Hypertension, Pulmonary; Connective Tissue Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Connective Tissue Diseases | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bosentan (Experimental)
  Interventions: Drug: bosentan

INTERVENTIONS:
Drug: bosentan — bosentan 62mg bid x 4 weeks, followed by bosentan 125mg bid x 20 weeks

SUMMARY:
The primary objectives of this exploratory study are to evaluate the effects of bosentan on hemodynamics (via cardiac catheterization) during exercise in patients with Pulmonary Arterial Hypertension (PAH) who have abnormal hemodynamics during exercise but normal hemodynamics at rest. The authors hypothesize that early treatment may change the course of disease progression by improving hemodynamics during exercise, thus delaying disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years of age
* For female patients, only non-pregnant women who are surgically sterile, postmenopausal or have documented infertility (over 50 years of age and amenorrheic for at least 1 year), or those of childbearing potential using one of the following methods of contraception:

  * Barrier-type devices (e.g., condom, diaphragm) used ONLY in combination with a spermicide. A double-barrier method is recommended.
  * Intrauterine devices (IUDs)
  * Oral contraceptives, if used in combination with a barrier method
* Body weight of 40 kg or higher
* Patients diagnosed with connective tissue disease
* Hemodynamics at rest, based on cardiac catheterization, should be as follows:

  * Mean pulmonary arterial pressure (mPAP) : 18 - 25 mmHg
  * PCWP ≤ 15 mmHg
* Hemodynamics during exercise, based on cardiac catheterization, should be as follows: mPAP > 30 mmHg
* Provide written informed consent

Exclusion Criteria:

* PAH associated with any other condition
* Severe obstructive lung disease : FEV1∕ FVC <0.5
* Total lung capacity <60% of normal predicted value
* Unable or unwilling have a cardiac catheterization procedure
* Acute or chronic impairment (other than dyspnea), limiting the ability to comply with study requirements (6-MWT)
* Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C
* AST and ∕or ALT > 3 times uln
* Hemoglobin concentration > 25% below the lower limit of normal
* Systolic blood pressure < 85 mm Hg
* Pregnancy or breast-feeding
* Treatment or planned treatment with another investigational drug
* Treatment with an endothelin receptor antagonist, phosphodiesterase type 5 inhibitor, or with prostanoids (excluding acute administration during a catheterization procedure to test vascular reactivity) within 2 months of inclusion
* Treatment with calcineurin-inhibitors (i.e., cyclosporine A and tacrolimus), fluconazole, glibenclamide (glyburide) within 1 week of study start;
* Known hypersensitivity to bosentan or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the change in the following hemodynamics during exercise: pulmonary vascular resistance (PVR), mean pulmonary arterial pressure (mPAP), cardiac output∕cardiac input (CO∕CI), mean right arterial pressure (mRAP) | 6 months

SECONDARY OUTCOMES:
Change in hemodynamics at rest: pulmonary vascular resistance (PVR), mean pulmonary arterial pressure (mPAP), cardiac output/cardiac input (CO∕CI), mean right arterial pressure (mRAP) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bradley, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Victoria Medical Center, Hamilton, Ontario, Canada